CLINICAL TRIAL: NCT03400579
Title: A Pilot Study of the Feasibility of Prehospital Delivery of Remote Ischemic Conditioning by Emergency Medical Services in Chest Pain Patients
Brief Title: A Study of the Feasibility of Prehospital Remote Ischemic Conditioning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 17-0287; UL1TR001111 (NIH)
Record Dates: First submitted 2018-01-08; First posted 2018-01-17 (Actual); Results first posted 2020-09-01 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2019-11

CONDITIONS: Chest Pain
Keywords: Emergency Medical Services
MeSH Terms: conditions — Chest Pain

STUDY DESIGN:
Intervention Model Description: Prospective, single center, single arm pilot study evaluating the feasibility of delivering remote ischemic conditioning by emergency medical services during ground ambulance transport of patients experiencing chest pain or anginal equivalent symptom
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Remote Ischemic Conditioning (Experimental): RIC procedure (i.e., four cycles of alternating 5-min inflation and 5-min deflation) administered by the autoRIC® device
  Interventions: Device: autoRIC® device

INTERVENTIONS:
Device: autoRIC® device — The autoRIC® automatically delivers four RIC cycles of five minutes of pressure at 200 mm Hg followed by five minutes of no pressure for a total 40-min treatment period

SUMMARY:
Prospective, single center, single arm pilot study evaluating the feasibility of delivering remote ischemic conditioning (RIC) by emergency medical services (EMS) in the prehospital setting. Eligible patients will have chest pain or anginal equivalent symptoms and require ground ambulance transport to the hospital. All subjects will undergo the standard RIC procedure (i.e., up to four cycles of alternating 5-min inflation and 5-min deflation) with the autoRIC® device (CellAegis Devices, Inc., Toronto, Ontario). The primary objective is to evaluate the number of cycles of RIC completed in patients having the procedure initiated by EMS in the prehospital setting.

DETAILED DESCRIPTION:
This single-arm, open-label pilot study will evaluate the feasibility of delivering remote ischemic conditioning (RIC) by emergency medical services (EMS) in the prehospital setting. Eligible patients will be at least 18 years of age, and require ground ambulance transport to the hospital. Patients suspected of ST-elevation myocardial infarction (STEMI) based on the prehospital electrocardiogram and thus requiring urgent intervention in the cardiac catheterization lab will be excluded.

All subjects will undergo the standard RIC procedure (i.e., up to four cycles of alternating 5-min inflation and 5-min deflation) with the autoRIC® device (CellAegis Devices, Inc.). The automated procedure will be initiated by paramedics during ambulance transport, and the RIC cycles will continue through emergency department (ED) arrival and stay for a total of 40 minutes.

The primary objective of this pilot study is to examine the duration of RIC administered in patients having the procedure initiated in the prehospital setting. The investigators hypothesize four cycles of RIC will be completed in at least 80% of patients having the procedure initiated. Secondary objectives are to assess enrollment rates and protocol implementation; paramedic acceptability of protocol; and patient tolerability of RIC.

ELIGIBILITY:
Inclusion Criteria:

1. Requiring 9-1-1 response to scene
2. At least 18 years of age
3. Experiencing non-traumatic chest pain or anginal equivalent symptom
4. Not meeting EMS criteria for a suspected STEMI based on prehospital ECG
5. Systolic blood pressure (SBP) between 100-180 mgm Hg
6. Designated for ambulance transport to University of North Carolina Medical Center (Chapel Hill, NC)
7. Capable of providing informed consent

Exclusion Criteria:

1. Unconscious or otherwise in critical condition
2. Lacking capacity to consent to the study
3. Non-English speaking
4. Pre-existing condition precluding blood pressure check or use of the autoRIC® at the discretion of the provider or listed here:

   1. Paresis of upper limb
   2. Pre-existing traumatic injury to arm
   3. Presence of an arteriovenous shunt for dialysis
   4. Prior mastectomy
   5. Existing peripheral inserted central catheter line
   6. Arm edema or other indication of upper extremity thrombosis
5. Serial ECG evidence of evolving STEMI

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mehul D Patel, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
The researchers have no plans to make individual participant data available. Due to this study's small size and single site, individual level data will not be shared to protect the privacy of subjects and maintain the confidentiality of data. Aggregated data and results on primary and secondary outcomes will be reported on this site and published in the scientific literature.

REFERENCES:
- [Derived] Patel MD, Platts-Mills TF, Grover JM, Thomas SM, Rossi JS. Feasibility of prehospital delivery of remote ischemic conditioning by emergency medical services in chest pain patients: protocol for a pilot study. Pilot Feasibility Stud. 2019 Mar 13;5:42. doi: 10.1186/s40814-019-0431-8. eCollection 2019. PMID 30911405

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Remote Ischemic Conditioning
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Remote Ischemic Conditioning
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 1
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10
Systolic Blood Pressure (mmHg) [Count of Participants; unit: Participants]
  100-120 | 3
  121-140 | 2
  141-160 | 4
  161-180 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects Receiving 4 Cycles of RIC Without Interruption
Description: A completed RIC cycle without interruption is defined as 5 minutes inflation followed by 5 minutes deflation for a total of 10 minutes.
Time Frame: up to 40 minutes, following initiation of RIC
Measure: Number; unit: percentage of participants
Arm/Group | Remote Ischemic Conditioning
Number analyzed (Participants) | 10
percentage of participants | 80

2. Secondary Outcome: Percent of Patients Screened Who Are Eligible for Recruitment
Description: Eligibility among patients screened and specifying inclusion and exclusion criteria met or not met.
Time Frame: through EMS transport, an average of 20 minutes
Population: Includes all patients screened for study eligibility
Measure: Number; unit: percentage of patients screened
Arm/Group | Remote Ischemic Conditioning
Number analyzed (Participants) | 11
percentage of patients screened | 100

3. Secondary Outcome: Percent of Patients Recruited Who Agreed to Participate
Description: Participation among patients who are screened and recruited.
Time Frame: through EMS transport, an average of 20 minutes
Population: Among all patients screened and determined to be eligible
Measure: Number; unit: percentage of patients recruited
Arm/Group | Remote Ischemic Conditioning
Number analyzed (Participants) | 11
percentage of patients recruited | 91

4. Secondary Outcome: Timing (in Minutes) of Study Procedures
Description: Times will be reported for on-scene arrival, patient transport, screening, recruitment, and RIC initiation to assess efficiency with which the study protocol was implemented. Screening, recruitment and RIC initiation times are overlapping with transport time.
Time Frame: through EMS response and transport, an average of 30 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Remote Ischemic Conditioning
Number analyzed (Participants) | 10
minutes
  On-Scene Time | 22.5 (5.6)
  Screening Time | 9.4 (10.0)
  Recruitment and RIC Start Time | 4.4 (8.7)
  Transport Time | 9.2 (4.6)

5. Secondary Outcome: Themes on Paramedic Acceptability of the Study Protocol
Description: Qualitative themes related to implementation of the study protocol will be derived from semi-structured interviews with study paramedics.
Time Frame: up to 15 minutes from screening
Population: The overall number of participants analyzed reflects participants undergoing the intervention (i.e., "Remote Ischemic Conditioning"). The study paramedics administering the intervention were not considered enrolled but contributed data for this assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Remote Ischemic Conditioning
Number analyzed (Participants) | 10
Participants
  Not enough time | 4
  Difficult to size the cuff | 4
  Ongoing training needed | 3

6. Secondary Outcome: Percent of Participants Experiencing Anticipated Adverse Events Including RIC Discontinuation Due to Discomfort
Description: Anticipated adverse events related to RIC including minor arm discomfort, temporary discoloration of the arm or hand, and minor skin bruising or abrasions on the upper arm will be collected via in-person and telephone evaluation.
Time Frame: up to 48 hours from end of RIC
Measure: Number; unit: percentage of participants
Arm/Group | Remote Ischemic Conditioning
Number analyzed (Participants) | 10
percentage of participants | 0

7. Secondary Outcome: Themes on Patient Experiences While Undergoing RIC
Description: Qualitative themes related to the RIC procedure will be derived from semi-structured interviews with subjects.
Time Frame: up to 15 minutes
Population: Includes participants that completed at least two RIC cycles
Measure: Count of Participants; unit: Participants
Arm/Group | Remote Ischemic Conditioning
Number analyzed (Participants) | 9
Participants
  Felt like a blood pressure cuff | 5
  Felt tight | 4

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of enrollment through 48 hours after.
Arm/Group | Remote Ischemic Conditioning
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-06-14): https://cdn.clinicaltrials.gov/large-docs/79/NCT03400579/Prot_SAP_ICF_001.pdf